CLINICAL TRIAL: NCT00741468
Title: An Open-Label, Multiple-Dose, Non-Randomized Study to Assess the Drug-Drug Interactions of Proellex® (CDB-4124) With Cytochrome P450 Isoenzymes CYP1A2, 2C9, 2C19, 2D6, and 3A4 in Healthy Female Subjects
Brief Title: Open-Label, Multiple-Dose, Non-Randomized Study to Assess Drug-Drug Interactions of Proellex® in Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZP-007
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Drug Interactions
Keywords: Drug-drug interactions; DDI
MeSH Terms: interventions — telapristone acetate; Caffeine; Tolbutamide; Omeprazole; Dextromethorphan; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Experimental): Proellex 50 mg CYP1A2 probe CYP2C9 probe CYP2C19 probe CYP2D6 probe CYP3A4 probe
  Interventions: Drug: Proellex; Drug: CYP1A2 probe; Drug: CYP2C9 probe; Drug: CYP2C19 probe; Drug: CYP2D6 probe; Drug: CYP3A4 probe

INTERVENTIONS:
Drug: Proellex — 2, 25 mg Proellex capsules administered daily
  Other Names: Telapristone acetate
Drug: CYP1A2 probe — Caffeine (200 mg)
  Other Names: Caffeine (200 mg)
Drug: CYP2C9 probe — Tolbutamide (250 mg)
  Other Names: Tolbutamide (250 mg)
Drug: CYP2C19 probe — Omeprazole (20 mg)
  Other Names: Omeprazole (20 mg)
Drug: CYP2D6 probe — Dextromethorphan (30 mg)
  Other Names: Dextromethorphan (30 mg)
Drug: CYP3A4 probe — Midazolam (2mg)
  Other Names: Midazolam (2mg)

SUMMARY:
This study will assess possible drug-drug interactions with specific isoenzymes over a total study duration of 6-8 weeks. Blood samples collected pre and post-dose, and urine samples collected post dose will be analyzed.

DETAILED DESCRIPTION:
This is an open-label, multiple-dose, non-randomized study to assess the drug-drug interactions of Proellex® with cytochrome P450 isoenzymes in healthy female subjects. On Day 1, following an overnight fast and morning void of the bladder, subjects will be administered CYP probe drugs orally. Serial blood samples will be collected at pre-dose and post-dose. Subjects will be administered two Proellex® 25 mg capsules (50 mg total dose) at approximately 0800 hours on Day 2 and 0700 hours on Days 3 through 8. One hour after administration of Proellex® on Day 8, the five CYP probe drugs will be administered and blood and urine samples collected as on Day 1. Blood samples for the determination of plasma concentrations of CDB-4124 and its metabolite CDB-4453 will be collected at pre-dose (trough) on Days 6, 7, and 8 to determine if steady-state conditions have been achieved. Samples will also be collected on Day 8 at 1, 2, 8 and 24 hour after administration of Proellex® to determine the plasma concentrations of CDB-4124 and CDB-4453.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult females
* A body mass index between 18 and 30 kg/m2, inclusive
* Negative urine drug and alcohol screen .

Exclusion Criteria:

* Significant medical condition,
* Significant physical examination finding
* Clinical laboratory
* ECG abnormality
* CYP2D6 "poor metabolizer"

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Wiehle, PhD, Study Director — Repros Therapeutics Inc.
Locations (1):
- Clinical Research Center Advanced Biomedical Research Inc., Hackensack, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: CYP1A2, Day 8 relative to Day 1 AUC (caffeine probe) CYP2C19, Day 8 relative to Day 1 AUC (omeprazole probe) CYP 2C9, Day 8 relative to Day 1 AUC (tolbutamide probe) CYP2D6, Day 8 relative to Day 1 AUC (dextromethorphan probe) CYP3A4, Day 8 relative to Day 1 AUC (midazolam probe)
Period: Overall Study
Arm/Group | All Participants
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects enrolled
Groups:
- All Subjects: Proellex 50 mg
  Proellex: 2, 25 mg Proellex capsules administered daily
Arm/Group | All Subjects
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Plasma AUC Ratio of Day 1 and Day 8
Description: Assessment of the drug-drug interactions of Proellex® (CDB-4124) with cytochrome P450 isoenzymes CYP1A2, 2C9, 2C19, 2D6, and 3A4 in healthy female subjects administered 50 mg Proellex® once daily (QD). The Day 8 AUC was compared to the Day 1 AUC to determine inhibition.
  For CYP1A2 the plasma paraxanthine/caffeine MR ratio (metabolic ratio) was used. For CYP2D6 the MR ratio of dextromethorphan/dextrorphan was used.
Time Frame: 8 days
Population: One subject had concentrations of Proellex (CDB-4124 and CDB-4453) that were below the lower level of quantitation at all time points tested and was excluded from the pharmacokinetic analyses.
Measure: Mean (90% Confidence Interval); unit: Ratio of geometric means Day 8 to Day 1
Groups:
- CYP1A2: Day 8 relative to Day 1 AUC (caffeine probe)
- CYP2C9: Day 8 relative to Day 1 AUC (tolbutamide probe)
- CYP2C19: Day 8 relative to Day 1 AUC (omeprazole probe)
- CYP2D6: Day 8 relative to Day 1 AUC (dextromethorphan probe)
- CYP3A4: Day 8 relative to Day 1 AUC (midazolam probe)
Arm/Group | CYP1A2 | CYP2C9 | CYP2C19 | CYP2D6 | CYP3A4
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 17
Ratio of geometric means Day 8 to Day 1 | 1.093 [1.006 to 1.188] | 1.029 [0.960 to 1.103] | 1.104 [0.936 to 1.303] | 1.914 [1.463 to 2.504] | 2.245 [2.019 to 2.495]

ADVERSE EVENTS:
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 13/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=18)
Early menstruation (Reproductive system and breast disorders) | 5 (5)
Headache (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 5 (5)
Lower back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bilateral leg cramps (Musculoskeletal and connective tissue disorders) | 2 (2)
Loose stools (Gastrointestinal disorders) | 2 (2)
Vaginal spotting (Reproductive system and breast disorders) | 1 (1)
Bilateral foot cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Lower abdominal cramps (Gastrointestinal disorders) | 1 (1)
Menstrual cramps (Reproductive system and breast disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights